CLINICAL TRIAL: NCT05943340
Title: Effects of Proprioceptive Training on Shoulder's Muscle Mass After Distal Radius Fracture. Randomized Clinical Trial.
Brief Title: Shoulder Proprioceptive Training During Immobilization of the Wrist
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Leire Cruz-Gambero, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RaqCan83
Record Dates: First submitted 2023-06-21; First posted 2023-07-13 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Wrist Fractures; Shoulder Pain
Keywords: Proprioceptive exercises; Function
MeSH Terms: conditions — Wrist Fractures; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be anonymized with a number and randomized with a web program (random.org)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients that are undergoing immobilization period after a distal radius fracture.
- Experimental group (Experimental): Patients that are undergoing immobilization period after a distal radius fracture.
  Interventions: Other: Proprioceptive exercises

INTERVENTIONS:
Other: Proprioceptive exercises — Specific proprioceptive exercises for the shoulder that the patient has to do during the immobilization period.
  Arms: Experimental group

SUMMARY:
The goal of this randomized clinical trial is to compare how a program of proprioceptive exercises for the shoulder could influence in pain, functionality, quality of life and shoulder muscle overload in people that are undergoing a immobilization period after a wrist fracture. The main questions it aims to answer are:

* Study the relationship between shoulder muscle overload and shoulder pain.
* Evaluate the effect of a proprioceptive program on pain and patient's satisfaction.

Intervention will be:

* Control group: participants of this group are not going to receive any protocol of exercises during the immobilization period.
* Experimental group: participants of this group are going to receive a protocol of proprioceptive shoulder exercises to do during the immobilization period.

Researchers will compare control and experimental group to see if a implantation of a proprioceptive program for the shoulder has benefits on pain, function, quality of life and muscle overload.

DETAILED DESCRIPTION:
Distal radius fracture (DRF) in one of the most frequent injuries in the upper limb, corresponding to 1/6 of the total fractures of the body. It appears mostly in >50 years old women (due to osteoporosis and menopause) but it is also frequent in middle age men as a consequence of a big trauma during sport activities or working. This injury can be treated conservative of surgically, but regardless of the treatment, it always has a period of immobilization between 3 to 6 weeks.

During the immobilization period, proximal structures suffer changes in mobility. Shoulder's ROM has to increased in order to compensate the immobilization of the wrist. Previous studies shown that there is a relation between time of immobilization and shoulder pain.

Shoulder pain can significantly affect daily living activities as driving, dressing or even eating. Also, pain does not appear only on it's own, but with other psychological factors as catastrophism, lower self-efficacy, fear of movement and avoidance. These factors could be crucial to predict disability in these patients, hence they should not be ignored during the rehabilitation process.

Our hypothesis is that the implementation of a proprioceptive shoulder exercise program during the period of immobilization may help and/or prevent shoulder pain secondary to immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Adult (equal or more than 18 y/o).
* Suffering a distal radius fracture and being in the first week of the immobilization period.
* Agree and sign informed consent.

Exclusion Criteria:

* Not had suffered a distal radius fracture and/or not being on the immobilization period.
* Suffer any mental, cognitive, neurological or musculoskeletal disorder.
* Previous injury or pathology of the shoulder diagnosed as fractures, instability, shoulder pain or capsulitis.
* Previous shoulder surgery.
* Have cervical pathology/impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-07-27 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in function related with daily living activities | Begining of the injury, baseline, 4 weeks and 3 months
  Measured with QuickDash. 11 items, 0= no disability and 100=total disability
Change in disability related with shoulder | Begining of the injury, baseline, 4 weeks and 3 months
  Measured with Shoulder Pain and Disability Index (SPADI). 13 items, with 2 subscales (pain and disability). Pain subscale goes from 0-50 points and disability subscale goes from 0 to 80 points. Total punctuation is expressed as a percentage. More points indicates more disability.
Change in perception of Pain, referred to shoulder | Begining of the injury, baseline, 4 weeks and 3 months
  Pain measured with Numerical Rating Scale (NRS). 0= no pain and 10=worst pain.

SECONDARY OUTCOMES:
Change in range of motion of the shoulder | Begining of the injury, baseline, 4 weeks and 3 months
  Active range of motion of the shoulder in all planes of motion
Change in Perception of Quality of life | Begining of the injury, baseline, 4 weeks and 3 months
  EuroQol-5D. It has 5 dimensions, mobility, self-care, daily activities, pain and anxiety and depression. Patient determines the level of agreement with the affirmations (3 options).
Change in shoulders muscle load | Begining of the injury, baseline, 4 weeks and 3 months
  Electromyographic study of the shoulder's muscles
Changes in catastrophizing pain | Begining of the injury, baseline, 4 weeks and 3 months
  Measured with Pain Catastrophizing Scale (PCS).13 items. Total punctuation goes from 0 to 52, where more points means more catastrophism level.
Changes in kinesiophobia, fear of movement | Begining of the injury, baseline, 4 weeks and 3 months
  Measured with Tampa Scale for Kinesiophobia (TSK). Punctuation goes from 17 to 68, from 36 points means presence of kinesiophobia.
Changes in fear of movement | Begining of the injury, baseline, 4 weeks and 3 months
  Measured with "Fear Avoidance Beliefs Q questionnarie" (FAB). 16 ítems. Punctuation goes from 0 to 96 points. More points means more fear and avoidance.
Changes in self-efficacy related to pain | Begining of the injury, baseline, 4 weeks and 3 months
  Measured with Chronic Pain Self-efficacy Scale (CPSES). 19 items. Punctuation goes from 0 to 60 points. High scores indicate greater levels of confidence in dealing with pain.